CLINICAL TRIAL: NCT07197450
Title: Efficacy and Safety of mRNA Drug XH02 in the Treatment of Adult Hypoparathyroidism
Brief Title: Efficacy and Safety of XH02 for the Treatment of Hypoparathyroidism
Acronym: XH02
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: K6744
Record Dates: First submitted 2025-09-14; First posted 2025-09-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hypoparathyroidism
Keywords: hypoparathyroidism; PTH; mRNA
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Intervention Model Description: accelerated titration combined with a 3+3 design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 20ug (Experimental): PTH1-84 mRNA 20ug
  Interventions: Drug: intravenous administration of PTH1-84 mRNA
- 40ug (Experimental): PTH1-84 mRNA 40ug
  Interventions: Drug: intravenous administration of PTH1-84 mRNA
- 80ug (Experimental): PTH1-84 mRNA 80ug
  Interventions: Drug: intravenous administration of PTH1-84 mRNA
- 120ug (Experimental): PTH1-84 mRNA 120ug
  Interventions: Drug: intravenous administration of PTH1-84 mRNA
- 160ug (Experimental): PTH1-84 mRNA 160ug
  Interventions: Drug: intravenous administration of PTH1-84 mRNA

INTERVENTIONS:
Drug: intravenous administration of PTH1-84 mRNA — intravenous administration of PTH1-84 mRNA

SUMMARY:
This study aims to evaluate the safety and efficacy of a novel PTH replacement therapy drug in patients with hypoparathyroidism. The drug is an mRNA drug which will be translated into PTH after intravenous administration, to achieve the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years (inclusive), male or female.
* Documented history of post-surgical chronic HP or autoimmune, genetic, or idiopathic HP for at least 26 weeks. Diagnosis of HP is confirmed based on a history of hypocalcemia accompanied by an inappropriately low serum PTH level (below the upper limit of the normal range of the local laboratory). * Note: If a subject lacks documented diagnosis of chronic HP but has exhibited hypocalcemia accompanied by an inappropriately low serum PTH level for at least 26 weeks prior to screening, and is judged by the investigator to meet the diagnostic criteria for chronic HP, they will be considered eligible for this criterion.
* Poorly controlled or intolerant to conventional therapy (calcium and active vitamin D).
* Conventional therapy (including vitamin D or magnesium supplements, if applicable) can be optimized during the screening period to achieve the following target serum levels: 25(OH) Vitamin D level: 10 - 100 ng/mL (25 - 250 nmol/L, inclusive). Blood magnesium level: Within the normal range or slightly below, i.e., ≥ 1.3 mg/dL (≥ 0.53 mmol/L). Albumin-corrected serum calcium (sCa) level: Within the normal range or slightly below
* Body Mass Index (BMI) of 17 to 40 kg/m² (inclusive) at screening.
* If aged ≤ 25 years, radiological evidence of closed epiphyses based on X-ray of the non-dominant hand (wrist and palm).

Exclusion Criteria:

* Impaired PTH response (pseudohypoparathyroidism), characterized by PTH resistance and elevated PTH levels in the presence of hypocalcemia.
* History of allergic predisposition, or known allergy to the investigational drug or polyethylene glycol (PEG)-containing medications.
* Any disease other than HP that may affect calcium metabolism, calcium-phosphate homeostasis, or PTH levels, such as: active hyperthyroidism; Paget's disease of bone; severe hypomagnesemia; type 1 diabetes mellitus or poorly controlled type 2 diabetes (HbA1c >9%; HbA1c results from within 12 weeks prior to screening are acceptable); severe and chronic liver or kidney disease; Cushing's syndrome; multiple myeloma; active pancreatitis; malnutrition; rickets; recent prolonged immobilization; active malignancy (except for low-risk, well-differentiated thyroid cancer or non-melanoma skin cancer); active hyperparathyroidism; history of parathyroid carcinoma within 5 years prior to screening; acromegaly; or multiple endocrine neoplasia syndromes.
* History of vaccination within 4 weeks prior to enrollment, or planned vaccination during the study period.
* Pregnant or lactating women.
* Patients with high-risk thyroid cancer requiring TSH suppression <0.2 mIU/L within the past 2 years, or patients with a history of malignancy.
* Requirement for long-term use of the following medications: diuretics, phosphate binders (except calcium supplements), digoxin, lithium, methotrexate, biotin >30 μg/day, or systemic corticosteroids (except as replacement therapy). Patients requiring long-term use of hormones or immunosuppressants (e.g., for rheumatologic/autoimmune diseases) are excluded. *Note: Subjects who can discontinue these medications for the study may be enrolled, provided the medications are stopped for at least 5.5 half-lives prior to blood sampling at Visit 1. Biotin must be stopped for at least 1 day prior to blood sampling during the screening period. These medications are prohibited throughout the entire study.*
* Use of PTH-like drugs (whether commercially available or obtained through participation in a clinical trial), including PTH(1-84), PTH(1-34), other N-terminal fragments or analogs of PTH, or PTH-related protein, within 4 weeks prior to screening.
* Participation in any other interventional trial involving an investigational drug or device within 8 weeks prior to screening, or within 5.5 half-lives of the administered drug from the previous trial (whichever is longer).
* Uncontrolled hypertension at baseline, OR a history of the following cardiovascular and cerebrovascular diseases: (1) Unstable angina; (2) Drug-requiring or severe arrhythmia; (3) Myocardial infarction; (4) Class III or higher heart failure (NYHA classification), or second-degree or higher atrioventricular block; (5) Cerebral infarction (except lacunar infarction), cerebral hemorrhage, or related diseases.
* Increased risk of osteosarcoma, such as Paget's disease of bone or unexplained elevated alkaline phosphatase; hereditary disorders predisposing to osteosarcoma; or patients who have received extensive external beam radiation therapy or implant radiation involving the skeleton.
* Clinically significant abnormal laboratory findings at screening, including any of the following:

Hematology: Neutrophil count (NEUT#) <1.5 × 10⁹/L; Platelet count (PLT) <90 × 10⁹/L; Hemoglobin (Hb) <90 g/L; Eosinophil count (EOS#) >0.5 × 10⁹/L.

Liver and Renal Function: Total bilirubin, Alanine Aminotransferase (ALT), or Aspartate Aminotransferase (AST) above the normal range; estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m².

* Any medical or other condition that, in the judgment of the Investigator, may affect the conduct of the study, interfere with the interpretation of study results, or pose an increased risk to the subject or the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
AE and SAE | the whole study period including the screening, treatment, and follow-up period. Follow-up period extends to 90 days after administration.
  adverse event (AE) and severe adverse event (SAE) via regular vital sign checks， physical examinations, and safety laboratory tests (including complete blood count, blood biochemistry, coagulation profile, C-reactive protein, urinalysis, cardiac ultrasound, and electrocardiogram).

SECONDARY OUTCOMES:
PTH1-84 | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  serum PTH1-84
PTH | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  serum PTH
serum calcium | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  serum calcium
Serum magnesium | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  Serum magnesium
Serum phosphorus | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  Serum phosphorus
1,25-dihydroxyvitamin D | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  serum 1,25-dihydroxyvitamin D
Fractional excretion of calcium （FECa) | Before (within 1 hour) and 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  FECa (%) = (Urine Calcium × Serum Creatinine) / (Serum Calcium × Urine Creatinine) × 100
24-hour urinary calcium | Before (within 3 days) and 24 hours, 48 hours, 72 hours after administration
  24-hour urinary calcium
Procollagen type I N-terminal propeptide (P1NP) | Before (within 1 hour) and 24 hours, 48 hours, 72 hours after administration
  serum procollagen type I N-terminal propeptide (P1NP)
Type I collagen cross-linked C-telopeptide (β-CTX） | Before (within 1 hour) and 24 hours, 48 hours, 72 hours after administration
  serum type I collagen cross-linked C-telopeptide (β-CTX）

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No